CLINICAL TRIAL: NCT03737188
Title: Institut Fuer Diabetes-Technologie Surveillance Program for Blood Glucose Monitoring Systems in Europe
Brief Title: Institut Fuer Diabetes-Technologie Surveillance Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDT-1722-IU
Record Dates: First submitted 2018-10-05; First posted 2018-11-09 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood glucose monitoring systems for self-testing — Capillary blood samples will be used for the evaluation of system accuracy.
  Other Names: 18 BGMS from 18 different manufacturers: ABRA, Accu-Chek Guide, AURUM Blutzucker-Messsystem, CareSens Dual, CERA-CHEK 1 Code, Contour next ONE, eBsensor, FreeStyle Freedom Lite, GL 50 (evo); GlucoCheck GOLD, GlucoMen areo 2K, GluNEO, MyStar DoseCoach, OneTouch Verio Flex, Pic GlucoTest, Rightest GM700S, TRUEyou Blutzuckermesssystem, WaveSense JAZZ WIRELESS

SUMMARY:
Assessment of the system accuracy of different blood glucose monitoring systems available in Europe

DETAILED DESCRIPTION:
A variety of blood glucose monitoring systems (BGMS) are available on the European market. For many of these BGMS, the system accuracy is unknown or it has not yet been assessed in manufacturer-independent studies. The IDT surveillance program aims at assessing the system accuracy of different BGMS that are available in Europe in a manufacturer-independent, investigator-initiated study. The initial study will cover 18 BGMS from 18 different manufacturers. Per BGMS, one test strip lot will be assessed based on procedures stated in the international standard ISO 15197:2013 / EN ISO 15197:2015.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or subjects without diabetes
* Signed informed consent form
* Minimum age of 18 years
* ubjects are legally competent and capable to understand character, meaning and consequences of the study.
* If blood glucose values < 80 mg/dl or > 300 mg/dl shall be measured after short term alteration in insulin therapy:
* Male or female with type 1 diabetes and intensified insulin therapy or insulin pump therapy.
* Signature of subjects to document consent with these procedures on informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Being unable to give informed consent
* < 18 years
* Legally incompetent
* Being committed to an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent on investigator or sponsor
* If blood glucose values < 80 mg/dl shall be measured after short term alteration in insulin therapy, subjects with type 1 diabetes, suffering from:
* Coronary heart disease
* Condition after myocardial infarction
* Condition after cerebral events
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on ISO 15197 | For each subject, the experimental phase has an expected duration of up to 6 hours
  Assessment of the analytical measurement performance of 18 blood glucose montoring systems based on procedures defined in ISO 15197

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Derived] Pleus S, Baumstark A, Jendrike N, Mende J, Link M, Zschornack E, Haug C, Freckmann G. System accuracy evaluation of 18 CE-marked current-generation blood glucose monitoring systems based on EN ISO 15197:2015. BMJ Open Diabetes Res Care. 2020 Jan;8(1):e001067. doi: 10.1136/bmjdrc-2019-001067. PMID 31958308